CLINICAL TRIAL: NCT04155840
Title: MRD-Guided Abbreviation of Bendamustine and Rituximab Chemotherapy in Combination With Copanlisib in Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Bendamustine and Rituximab in Combination With Copanlisib for the Treatment of Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: University of Washington (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Ryan Lynch, Assistant Professor, Division of Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005103; NCI-2019-07289 (Registry Identifier: NCI / CTRP); 10325 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Results first posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Lymphoid Leukemia; Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphoid; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — copanlisib; Rituximab; CT-P10; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (copanlisib, rituximab, bendamustine) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8 and 15 or days 1 and 15 (depending on dose level). Patients also receive rituximab IV on day 1 and bendamustine IV on days 1 and 2 of cycles 1-4. Patients who achieve at least a partial response (MRD-positive) continue on treatment for 2 additional cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 7, patients receive copanlisib IV over 1 hour on days 1 and 15 for an additional 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Biological: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: Copanlisib — Given IV
  Other Names: 1032568-63-0; BAY 80-6946; PI3K Inhibitor BAY 80-6946
Biological: Rituximab — Given IV
  Other Names: C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar GB241; Rituximab Biosimilar JHL1101; Rituximab Biosimilar SAIT101; RTXM83; Truxima
Drug: Bendamustine — Given IV
  Other Names: 16506-27-7; SDX-105

SUMMARY:
This trial studies how well bendamustine and rituximab in combination with copanlisib work in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma. Drugs used in chemotherapy, such as bendamustine and rituximab, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Copanlisib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving bendamustine and rituximab with copanlisib may work better than bendamustine and rituximab alone in treating chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
This is a dose de-escalation study of copanlisib.

Patients receive copanlisib intravenously (IV) over 1 hour on days 1, 8, and 15 or days 1 and 15 (depending on dose level). Patients also receive rituximab IV on day 1 and bendamustine IV on days 1 and 2 of cycles 1-4. Patients who achieve at least a partial response (MRD-positive) continue on treatment for 2 additional cycles. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Beginning cycle 7, patients receive copanlisib IV over 1 hour on days 1 and 15 for an additional 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 14 days, then periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, non-17p del chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) with any of the three following conditions:

  * No prior CLL/SLL directed therapy and Cumulative Illness Rating Scale (CIRS) score >= 7
  * Age >= 65
  * At least one prior CLL/SLL directed therapy with any CIRS score
* CLL/SLL requiring treatment as defined by at least one of the following criteria based on IWCLL 2018 guidelines:

  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
  * Massive (> 6 cm below left costal margin), progressive or symptomatic splenomegaly
  * Massive nodes (> 10 cm in longest diameter), or progressive or symptomatic lymphadenopathy
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period or lymphocyte-doubling time of < 6 months. Lymphocyte-doubling time may be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In patients with initial blood lymphocyte counts of < 30x10^9/L (30,000/uL), lymphocyte-doubling time should not be used as a single parameter to define treatment indication. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL/SLL (eg, infection, steroid administration) should be excluded
  * Constitutional symptoms, defined as any 1 or more of the following disease-related symptoms or signs:

    * Unintentional weight loss of > 10% within the previous 6 months
    * Significant fatigue (ie, inability to work or perform usual activities)
    * Fevers > 100.5 degrees Fahrenheit (F) or 38 degrees Celsius (C) for? 2 weeks without other evidence of infection
  * Night sweats for > 1 month without evidence of infection
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Previous exposure to other PI3K inhibitors (except copanlisib) is acceptable provided there is no resistance (resistance defined as no response [response defined as partial response (PR) or complete response (CR)]) at any time during therapy, or progressive disease (PD) after any response (PR/CR) or after stable disease within 6 months from the end of the therapy with a PI3K inhibitor
* Willingness and ability to comply with study and follow-up procedures, and give written informed consent
* Female subjects of childbearing potential must be surgically sterile, be post-menopausal (per institutional guidelines), or must have a negative serum pregnancy test within 7 days prior to cycle 1 day 1 and agree to use medically acceptable contraception throughout the study period and for 4 months after the last dose of either study drug. Men of reproductive potential may not participate unless they agree to use medically acceptable contraception throughout the study period and for 4 months after the last dose of either study drug
* Patients must be expected to receive at least 2 cycles of therapy
* Patients should have an expected survival if untreated of >= 90 days
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (< 3 x ULN for patients with Gilbert-Meulengracht syndrome or for patients with cholestasis due to compressive adenopathies of the hepatic hilum) (collected no more than 7 days before starting study treatment)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement by lymphoma) (no more than 7 days before starting study treatment)
* Lipase =< 1.5 x ULN (no more than 7 days before starting study treatment)
* Glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2 according to the Modification of Diet in Renal Disease (MDRD) abbreviated formula (no more than 7 days before starting study treatment). If not on target, this evaluation may be repeated once after at least 24 hours either according to the MDRD abbreviated formula or by 24 hour sampling. If the later result is within acceptable range, it may be used to fulfill the inclusion criteria instead
* International normalized ratio (INR) =< 1.5 and partial thromboplastin time (PTT) =< 1.5 x ULN. Prothrombin time (PT) can be used instead of INR if =< 1.5 x ULN (collected no more than 7 days before starting study treatment)
* Platelet count >= 75,000 /mm^3. For patients with confirmed lymphomatous bone marrow infiltration, platelet count >= 50,000 /mm^3 (collected no more than 7 days before starting study treatment)
* Hemoglobin (Hb) >= 8 g/dL (collected no more than 7 days before starting study treatment). Packed red blood cell transfusion or erythropoietin should not be given less than 7 days before the exam collection
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (collected no more than 7 days before starting study treatment). For patients with confirmed lymphomatous bone marrow infiltration, ANC count >= 750/mm^3. Myeloid growth factors should not be given less than 7 days before the exam collection

Exclusion Criteria:

* Presence of chromosome 17p deletion, known p53 deletion, or known p53 mutation that impairs normal function
* Prior treatment including systemic therapy or radiotherapy within 21 days of study initiation
* Prior treatment with bendamustine within 2 years
* Prior treatment with copanlisib
* Documented evidence of resistance to prior treatment with idelalisib or other PI3K inhibitors defined as: No response (response defined as partial response [PR] or complete response [CR]) at any time during therapy, or Progression (PD) after any response (PR/CR) or after stable disease within 6 months from the end of the therapy with a PI3K inhibitor
* Active autoimmune disease or prior autoimmune disease requiring systemic immunosuppression within the past 6 months
* Poorly controlled diabetes mellitus defined as hemoglobin A1c > 8.5%
* Known lymphomatous involvement of the central nervous system
* Known history of human immunodeficiency virus (HIV) infection. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations
* Hepatitis B (hepatitis B virus [HBV]) or C (hepatitis C virus [HCV]) infection. All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel. Patients positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV-deoxyribonucleic acid (DNA), these patients should receive prophylactic antiviral therapy. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-ribonucleic acid (RNA)
* Previous or concurrent history of malignancies within 3 years prior to study. Any exceptions beyond those listed below must be approved by the principal investigator:

  * Cervical carcinoma in situ
  * Non-melanoma skin cancer
  * Superficial bladder cancer (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
  * Localized prostate cancer
* Active, clinically serious infections (> Common Terminology Criteria for Adverse Events [CTCAE] grade 2)
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Proteinuria of >= CTCAE grade 3 as assessed by a 24 hours (h) total urine protein quantification or estimated by urine protein : creatinine ratio > 3.5 on a random urine sample
* Unresolved toxicity from prior therapy higher than National Cancer Institute (NCI)-CTCAE grade 1 attributed to any prior therapy/procedure excluding alopecia or sensory neuropathy. Concurrent diagnosis of pheochromocytoma
* Pregnant or breast-feeding patients. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study result
* Congestive heart failure > New York Heart Association (NYHA) class 2
* Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
* Myocardial infarction less than 6 months before start of test drug
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's assessment)
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 3 months before the start of study treatment
* Non-healing wound, ulcer, or bone fracture
* Patients with seizure disorder requiring medication
* Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event >= CTCAE grade 3 within 4 weeks prior to the start of study treatment
* Any illness or medical conditions that are unstable or could jeopardize the safety of the patients and their compliance in the study
* History of having received an allogeneic bone marrow or organ transplant
* Anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Major surgical procedure or significant traumatic injury (as judged by the investigator) less than 28 days before start of treatment, open biopsy less than 7 days before start of treatment
* Systemic continuous corticosteroid therapy at a daily dose higher than 15 mg prednisone or equivalent is not allowed. Patients may be using topical or inhaled corticosteroids. Previous corticosteroid therapy must be stopped or reduced to the allowed dose at least 7 days performing the screening computed tomography (CT)/magnetic resonance imaging (MRI). If a patient is on chronic corticosteroid therapy, corticosteroids should be de-escalated to the maximum allowed dose before the screening. Patients may be using topical or inhaled corticosteroids
* Use of CYP3A4 inhibitors and inducers. Copanlisib is primarily metabolized by CYP3A4. Therefore, concomitant use of strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir), and strong inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) are not permitted from day -14 of cycle 1 until the end of treatment visit

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lynch, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 72 [72 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Estimate the Marrow Minimal Residual Disease (MRD)-Negative Rate
Description: Will use a Simon optimal two-stage design.
Time Frame: End of cycle 4 (each cycle is 28 days)
Population: Data for the outcome measure was collected, however, the outcome measure was not analyzed because we were unable to determine the marrow minimal residual disease (MRD)-negative rate due to low accrual and few data timepoints for which meaningful data could be extracted.
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Number analyzed (Participants) | 0

2. Secondary Outcome: Marrow MRD-negative Rate
Time Frame: At 1 year
Population: Data for the outcome measure was not collected.
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: At 1 and 3 years
Population: Data for the outcome measure was not collected.
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Number analyzed (Participants) | 0

4. Secondary Outcome: MRD Conversion Rate Among Those Who Are MRD-positive After 4 Cycles
Time Frame: End of cycle 4 (each cycle is 28 days)
Population: This outcome measure was not done. The MRD sample after Cycle 4 was received at the analyzing lab beyond stability.
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportion of Subjects Who Experience Grade 3+ Immune-mediated Adverse Events or Any Grade 5 Adverse Event Possibly Related to Copanlisib
Time Frame: Approximately 6 months
Population: Data for the outcome measure was collected, however, the outcome measure was not analyzed due to low accrual and few data timepoints for which meaningful data could be extracted.
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected after the first administration of copanlisib until the end of treatment visit, approximately 6 months.
Description: Adverse events are collected through regular investigator assessment, regular laboratory testing, and patient interviews.
Arm/Group | Treatment (Copanlisib, Rituximab, Bendamustine)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Copanlisib, Rituximab, Bendamustine) (N=1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Flatulance (Gastrointestinal disorders) | 1 (1)
Knots on forehead (General disorders) | 1 (1)
Bilateral nipple pain (General disorders) | 1 (2)
Gynecomastia (Reproductive system and breast disorders) | 1 (1)
Infusion-related reaction (Injury, poisoning and procedural complications) | 1 (5)
Bilateral ankle edema (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Clammy feeling (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (3)
Papule on back (Skin and subcutaneous tissue disorders) | 1 (1)
Flaking lesion, right cheek (Skin and subcutaneous tissue disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Low accrual precluded statistical analyses and other results analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT04155840/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04155840/ICF_000.pdf